CLINICAL TRIAL: NCT06970600
Title: Monitoring the Therapeutic Efficacy of Artemether-Lumefantrine Combination in the Treatment of Uncomplicated Plasmodium Falciparum Malaria in Children Under 12 Years of Age at Four Sentinel Sites in Mozambique
Brief Title: Efficacy of Artemether-Lumefantrine in the Treatment of Uncomplicated Plasmodium Falciparum Malaria in Children Under 12 Years at Four Sentinel Sites in Mozambique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro de Investigacao em Saude de Manhica (Other)
Collaborators: World Health Organization (Mozambique) (Unknown); National Malaria Control Program (NMCP), Mozambique (Unknown); Instituto Nacional de Saúde, Mozambique (Other Government)
Responsible Party: Principal Investigator, Pedro Aide, PhD, Centro de Investigacao em Saude de Manhica
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEFI_V; SUB CONTRACT AGREEMENT #1 (Other Grant/Funding Number: Medical Care Development Global health (MCD))
Record Dates: First submitted 2025-05-06; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Malaria (Uncomplicated)
Keywords: Efficacy; Artemether-lumefantrine; Mozambique; Malaria
MeSH Terms: conditions — Malaria | interventions — Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Artemether-lumefantrine (Other): AL (Coartem™) will be administered twice daily for three days (six doses in total) with dosage determined according to body weight: one tablet (20mg artemether and 120mg lumefantrine) for children 5 to <15kg, two tablets per dose for those 15 to <25kg, and three tablets per dose for those 25 to <35kg.
  Interventions: Drug: Artemether-lumefantrine (Coartem)

INTERVENTIONS:
Drug: Artemether-lumefantrine (Coartem) — Eligible patients will be consecutively assigned to the four cohorts. Rescue therapy according to national malaria treatment guidelines will be also administered in cases of early or late treatment failure. Follow-up visits will take place on days 1, 2, 3, 7, 14,21 and 28 after enrolment or at any time point whenever the child is sick. Adverse events will be recorded and assessed for severity and association with study medication. Thick and thin Giemsa-stained blood slides will be prepared before each dose to be administered and at every follow-up visit of days 2, 3, 7, 14, 21, 28, 35 and 42. Blood samples for PCR analysis will be collected from every patient at baseline and at days 7, 14, 28, and 42 day of treatment failure or at any other unscheduled visit. To differentiate recrudescence from new infection by polymerase chain reaction (PCR) analysis.The Molecular markers associated with suboptimal response to ACTs will be investigated.

SUMMARY:
This is a classical in vivo clinical trial, following World Health organization's recommendations, ran as a multisite study within Mozambique trying to assess the efficacy and safety in four sites of artemether-lumefantrine (AL) combination for the treatment of uncomplicated malaria in children aged<12 years. The goal of this study is to evaluate the clinical and parasitological efficacy of the study drug combinations in children aged between 6 - 143 months, suffering from uncomplicated P. falciparum malaria, by determining the proportion with early treatment failure (ETF), late clinical failure (LCF), late parasitological failure (LPF) or an adequate clinical and parasitological response (ACPR) as indicators of efficacy. The participants will take AL for three days and followed-up for 28 days.

DETAILED DESCRIPTION:
Eligible patients were consecutively assigned to the cohort and treated with AL. AL (Coartem™) will be administered twice daily for three days (six doses in total) with dosage determined according to body weight: one tablet (20mg artemether and 120mg lumefantrine) for children 5 to <15kg, two tablets per dose for those 15 to <25kg, and three tablets per dose for those 25 to <35kg. All treatments will be directly observed for a minimum of 30 minutes. Vomiting occurring within the first 30 minutes implied the repetition of the full dose of treatment. For those patients living far away from the health facilities, and for which direct observation of the evening doses of AL was challenging, admission was offered for the first three days of the study. Then after first four days, the patients were followed-up weekly ( clinical and laboratory assessment) until day 28.

ELIGIBILITY:
Inclusion Criteria:

* Ages 6 to 143 months
* Weight Greater than or equal to 5 kg
* Absence of severe malnutrition;
* Mono-infection with Plasmodium falciparum in blood, confirmed by microscopy;
* Parasite density between 1,000 and 200,000 asexual parasites per microliter of blood;
* Haemoglobin ≥ 7.0 g/dl;
* Axillary temperature ≥ 37.5 C° or history of fever in the last 24 hours;
* Lack of danger signs, or no signs of severe and / or complicated malaria according to the WHO definition
* Ability to swallow the drugs
* Residents within the study area and have the possibility of an adequate follow-up in the days of monitoring for a period of 28 days;
* Absence of a history of hypersensitivity to study medications;
* Informed consent of parents, guardians or caregivers (legal guardian) after explaining the purpose of the study.

Exclusion Criteria:

* Presence of any danger sign or severe or complicated Plasmodium falciparum malaria according to WHO definitions;
* Presence of fever due to diseases other than malaria (eg measles, acute respiratory infection, severe diarrhea with dehydration) or other known diseases, with chronic or serious illnesses (cardiac, renal, hepatic or known infection with HIV AIDS);
* Presence of severe malnutrition (defined as a child whose growth pattern is below the 3rd percentile, mid-upper-arm circumference <110mm, weight / height <70% according to the WHO tables, or the presence of bilateral edema of the lower limbs);
* Multi or mono-infection by another Plasmodium species detected by microscopy;
* Regular medication that may interfere with the pharmacokinetics of antimalarials;
* History of hypersensitivity or contraindication to study drug;
* A history of taking antimalarial drugs or drugs with antimalarial activity in less than 7 days.
* Continuous prophylaxis with cotrimoxazole in HIV positive children.

Ages: 6 Months to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 352 (Actual)
Dates: Start 2024-03-07 (Actual); Primary Completion 2024-10-28 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Measuring the Day 28, PCR corrected cure rates of artemether-lumefantrine. | 28 days
  This cure rate is defined as the proportion of patients with adequate clinical and parasitological response (ACPR) at Day 28, once PCR correction to differentiate recrudescences from new infections have been applied (and hence only considering as treatment failures those parasite recurrences confirmed as recrudescences).

SECONDARY OUTCOMES:
To evaluate the incidence of adverse events | 28 days
  Safety was assessed by administering a questionnaire about the nature and incidence of adverse events and serious adverse events. An adverse event is defined as any unfavorable, unintended sign, symptom, syndrome or disease that develops or worsens with the use of a medicinal product, regardless of whether it is related to the medicinal product.
To evaluate the variation of the levels of haemoglobin during and after treatment | 28 days
  Haemoglobin levels were measured on Day 0, Day 14 and Day 28 using a haemoglobinometer and their levels were compared at these three points.
Measuring the Day PCR uncorrected cure rates of Artemether-Lumefantrine. | 28 days
  This cure rate is defined as the proportion of patients with adequate clinical and parasitological response (ACPR) at Day 28, without PCR correction to differentiate recrudescences from new infections and hence considering as treatment failures all parasite recurrences.
Evaluate the presence of Molecular Markers associated with sub optimum responses to ACTs | 28 days
  The presence of molecular marks is defined as presence of mutations in pfk13 and pfmdr1 (at codons 86, 184 and 1246) genes identified by Sanger sequencing of pre-treatment samples.

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Aide, MD, Msc, PhD, Principal Investigator — Centro de Investigaçao em Saude de Manhiça
Locations (4):
- Mozambique (4):
  - Hospital Distrital de Massinga, Massinga, Inhambane Province
  - Hospital Rural de Cuamba, Cuamba, Niassa Province
  - Hospital Distrital de Dondo, Dondo, Sofala
  - Hospital Distrital de Mopeia, Mopeia, Zambezia Province

IPD SHARING:
Plan to Share IPD: Undecided